CLINICAL TRIAL: NCT02524132
Title: Physical Activity Intervention in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Hamline University (Unknown)
Responsible Party: Principal Investigator, James Levine, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0812015
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Activity (Experimental): 5 minute movement breaks
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity

SUMMARY:
In this research project, the investigators addressed if incorporating physical movements with preschoolers will help increase their ability to retain concepts learned in preschool such as letter, sound and number recognition. Movement plays an important role in the brain. Exercise shows many benefits for the brain to help maintain clearer thought, improve memory, and increase activity in the brain, especially the areas involved in memory, attention, and language. The following research includes an eight week study of the implementation of movement breaks with one preschool class, while using another class as a control group. During the two weeks of baseline data, data was collected from every student in both groups on their letter recognition with both upper and lower case, letter sound identification, and number recognition for numbers 0-10. The group that implemented movement breaks had three-five minute scheduled times to stop for movement. Data was collected and compared between the two groups to find differences in their academic performance.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled preschool student

Exclusion Criteria:

* Enrolled in multiple preschool classes

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Physical Activity as measured by a Modular Signal Recorder Accelerometer | 8 wks
Letter recognition as measured by an Academic Growth Assessment | 8 wks
Sound recognition as measured by an Academic Growth Assessment | 8 wks
Number recognition as measured by an Academic Growth Assessment | 8 wks

CONTACTS AND LOCATIONS:
Locations (1):
- Hamline University, Saint Paul, Minnesota, United States